CLINICAL TRIAL: NCT05601947
Title: Investigation of the Effectiveness of Wii-Based Exercise Play Therapy in Knee
Brief Title: Investigation of the Effectiveness of Wii-Based Exercise Play Therapy in Knee Osteoarthritis Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gulerbuyukyilmaz, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-65142
Record Dates: First submitted 2022-10-25; First posted 2022-11-01 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
Keywords: Virtual Reality; Exercise; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Proprioception and Closed Kinetic Chain Exercises Group (Experimental): In addition to electrotherapy and conventional exercise program applications, structured proprioception and closed kinetic chain exercises will be applied for 3 weeks under the supervision of a physiotherapist. A rest period of 10 seconds will be given between exercises.
  Interventions: Other: Structured Proprioception and Closed Kinetic Chain Exercises Group
- Wii Based Balance Training Program Group (Experimental): In addition to electrotherapy and conventional exercise program, wii-based balance training program will be applied 5 days a week for 3 weeks.
  Interventions: Other: Wii Based Balance Training Program Group

INTERVENTIONS:
Other: Structured Proprioception and Closed Kinetic Chain Exercises Group — In this group, an exercise program consisting of 3 stages, ranging from simple to difficult and including closed kinetic chain exercises and proprioceptive exercises, will be applied.
  Arms: Structured Proprioception and Closed Kinetic Chain Exercises Group
Other: Wii Based Balance Training Program Group — In addition to electrotherapy and conventional exercise program, wii-based balance training program will be applied 5 days a week for 3 weeks. "Balance Surf", which includes lateral weight transfer, "Balance Adventure", which includes versatile balance exercises, and "balance bowling" for static and dynamic postural control will be implemented in the Fizyosoft Balance System. Each game will be practiced under the supervision of a physiotherapist for a total of 3 minutes, respectively, Balance surf, Balance adventure, Balance surf, Balance bowling and Balance surf, for a total of 15 minutes.
  Arms: Wii Based Balance Training Program Group

SUMMARY:
Osteoarthritis (OA) is a slowly progressive, chronic and degenerative joint disease frequently seen in the knee and hip joints. OA is not only involved in degenerative changes of cartilage, but can also be a result of capsular hypertrophy, osteophytes, subchondral bone sclerosis, ulcerations, fibrillations. It progressively impairs the patient's independence, mobility and participation in social life, thus reducing the overall quality of life. Edema, stiffness, instability, decreased muscle strength, impaired range of motion and proprioceptive sensation, increased incidence of falls are seen together with the main symptom of pain. In OA, treatment options are available to manage symptoms and optimize quality of life. In clinical guidelines, evidence-based treatment for Osteoarthritis may include patient education and self-management programs that integrate weight management, structured exercise, and physical activity. Closed kinetic chain exercises have gained importance in the rehabilitation of many musculoskeletal problems in the last 20 years and have become one of the most preferred exercises. In addition, the virtual reality treatment approach, which is the most common example of technology use in rehabilitation, has also started to take place in rehabilitation studies. The aim of this project is to investigate the effects of Wii-based video-based exercise game therapy on muscle strength, proprioception, postural control and functional level in knee osteoarthritis rehabilitation.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a slowly progressive, chronic and degenerative joint disease frequently seen in the knee and hip joints. OA is not only involved in degenerative changes of cartilage, but can also be a result of capsular hypertrophy, osteophytes, subchondral bone sclerosis, ulcerations, fibrillations. It progressively impairs the patient's independence, mobility and participation in social life, thus reducing the overall quality of life. Edema, stiffness, instability, decreased muscle strength, impaired range of motion and proprioceptive sensation, increased incidence of falls are seen together with the main symptom of pain. In OA, treatment options are available to manage symptoms and optimize quality of life. In clinical guidelines, evidence-based treatment for Osteoarthritis may include patient education and self-management programs that integrate weight management, structured exercise, and physical activity. Closed kinetic chain exercises have gained importance in the rehabilitation of many musculoskeletal problems in the last 20 years and have become one of the most preferred exercises. In addition, the virtual reality treatment approach, which is the most common example of technology use in rehabilitation, has also started to take place in rehabilitation studies. The aim of this project is to investigate the effects of Wii-based video-based exercise game therapy on muscle strength, proprioception, postural control and functional level in knee osteoarthritis rehabilitation.

Method: 56 volunteers diagnosed with bilateral knee OA, who underwent routine electrotherapy and conventional exercise program in the laboratory of Istanbul Rumeli University and were directed to exercise according to the inclusion criteria, will be included in the study. Patients with knee pain due to OA for at least 6 months, diagnosed with primary OA according to the criteria of the American College of Rheumatology, Stage 2-3 knee OA according to the Kellgren-Lawrence classification, aged 55-65, without any neurological disease Individuals who volunteered to participate and had a Mini Mental State Scale score ≥23 will be included. Diagnosed with secondary OA, Operated on the knee, hip and/or spine, Severe knee trauma or physical therapy for the knee in the last year, Presence of neurological disease that may affect balance and proprioception, Vertigo, hearing and vision problems, Genu varum and Genu valgum and Individuals with scoliosis, Body Mass Index (BMI) ≥40 kg/m2 and Visual analog scale ≥8/10 will be excluded from the study. Pain with Visual Analog Scale, pain threshold with algometer, range of motion with goniometer, muscle strength with dynamometer, functional level with Western Ontario and McMaster Universities Osteoarthritis Index and Lequesne knee index, postural control with Berg balance scale, functional performance with timed get up and go test, 10 meters walking test and 10 steps climbing test, and proprioception with digital goniometer will be evaluated for all participants before and after treatment and at the 8th week of treatment. All individuals participating in the study will be randomly divided into 2 groups. All individuals participating in the study will receive 15 sessions of electrotherapy and conventional exercise program, 5 days a week for 3 weeks. In the first group, besides electrotherapy and conventional exercise program applications, structured proprioception and closed kinetic chain exercises will be applied for 3 weeks under the supervision of a physiotherapist. A rest period of 10 seconds will be given between exercises. The second group will be given a wii-based balance training program for 3 weeks, 5 days a week, in addition to the electrotherapy and conventional exercise program. It was aimed to find an effective treatment method in individuals with knee osteoarthritis by comparing the groups at the end of the treatment and at the 8th week.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee pain due to OA for at least 6 months,
* diagnosed with primary OA according to the criteria of the American College of Rheumatology,
* Stage 2-3 knee OA according to the Kellgren-Lawrence classification,
* aged 55-65,
* without any neurological disease
* Individuals who volunteered to participate
* Patients with a Mini Mental State Scale score ≥23

Exclusion Criteria:

* Diagnosed with secondary OA,
* Patients who have undergone surgery to the knee, hip and/or spine,
* Severe knee trauma
* Have had physical therapy for the knee in the past year
* Presence of neurological disease that may affect balance and proprioception,
* Vertigo, hearing and vision problems,
* Genu varum and Genu valgum and Individuals with scoliosis,
* Patients with a body Mass Index (BMI) ≥40 kg/m2
* Patients with a visual analog scale ≥8/10

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
VAS | 5 minutes
  The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
pain threshold | 5 minutes
  with algometer
Normal range of motion | 5 minutes
  Normal range of motion can be measured with goniometer
muscle strength | 5 minutes
  muscle strength is measured with a dynamometer
proprioception | 10 minutes
  digital goniometer
Evaluation of Functional Performance | 5 minutes
  Functional performance was evaluated with the Timed Up and Go Test
Evaluation of Functional Performance | 5 minutes
  Functional performance was evaluated with the 10-meter walk test
Evaluation of Functional Performance | 5 minutes
  Functional performance was evaluated with the 10-step climbing test.

SECONDARY OUTCOMES:
functional level | 10 minutes
  Western Ontario and McMaster Universities Osteoarthritis Index
functional level | 10 minutes
  lequesne knee index
postural control | 10 minutes
  The Berg Balance Scale (BBS) consists of 14 different questions that evaluate the maintenance of the static position during changes in the orientation of the body center of gravity. Scoring is made between 0-4. In this scoring, 4 points represent the activity without any support, while 0 points represent full support or not performing the activity at all. The highest total score is 56 and reflects perfect balance.If the patient scores between 0-20 points, she is considered wheelchair dependent.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will publish my manuscript about this study, so researchers can access my individual participant data with this way.

REFERENCES:
- [Result] Manlapaz DG, Sole G, Jayakaran P, Chapple CM. Exergaming to improve balance and decrease the risk of falling in adults with knee osteoarthritis: a mixed-methods feasibility study. Physiother Theory Pract. 2022 Nov;38(13):2428-2440. doi: 10.1080/09593985.2021.1952670. Epub 2021 Jul 19. PMID 34280069